CLINICAL TRIAL: NCT01867021
Title: A Multi-Center, Phase IV, Randomized, Controlled, Observer Blind Study to Evaluate the Immunogenicity, Safety, and Tolerability of a Trivalent Subunit Inactivated Influenza Vaccine in Healthy Subjects Aged 50 Years and Above
Brief Title: Immunogenicity, Safety and Tolerability of a Trivalent Subunit Inactivated Vaccine in Healthy Subjects 50 Years and Above
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V71_22
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Influenza
Keywords: Trivalent inactivated subunit influenza vaccines; 50 years and above; healthy subjects
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agriflu (Experimental): A single 0.5 mL dose of Investigational vaccine TIV (Agriflu) at visit 1, administered intramuscularly
  Interventions: Biological: Agriflu (TIV)
- Fluvirin (Active Comparator): A single 0.5 mL dose of control vaccine TIVf (Fluvirin) at visit 1, administered intramuscularly
  Interventions: Biological: Fluvirin(TIVf)

INTERVENTIONS:
Biological: Fluvirin(TIVf)
  Other Names: Trivalent Influenza Virus Vaccine (purified surface antigen, inactivated, egg-derived)
  Arms: Fluvirin
Biological: Agriflu (TIV)
  Other Names: Trivalent Influenza Virus Vaccine (purified surface antigen, inactivated, egg-derived)
  Arms: Agriflu

SUMMARY:
Demonstrate non-inferiority of the post-vaccination (Day 22) Hemagglutination inhibition (HI) Geometric Mean Titers (GMTs) of trivalent, inactivated, subunit influenza vaccine (TIV) over the corresponding GMTs of the comparator vaccine for all three strains, in healthy adults aged 50 years and above.

Demonstrate non-inferiority of the percentages of subjects achieving seroconversion in antibody titers at Day 22 in the TIV group over the corresponding percentages of subjects in the comparator group for all three strains, in healthy adults aged 50 years and above.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 50 years and above, mentally competent, willing and able to give written informed consent prior to study entry and after the nature of the study has been explained according to local regulatory requirements.
* Individuals able to comply with all the study requirements.
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
* Individuals with any progressive or severe neurologic disorder, seizure disorder or Guillain-Barré syndrome.
* Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study.
* Individuals who have received any seasonal or pandemic influenza vaccine or have had a laboratory confirmed seasonal or pandemic influenza disease within the past 6 months.
* Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
* Individuals with positive HIV test result, with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy within 6 months or use of any parenteral or oral corticosteroids within the previous 30 days.
* Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Individuals with any serious chronic or progressive disease according to judgment of the investigator (neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
* Individuals who have any malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder.
* Individuals with history of any anaphylactic adverse event and/or serious allergic adverse event following a vaccination, a proven hypersensitivity to any component of the study vaccine (eg, to eggs or eggs product as well as ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate) or latex allergy.
* Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
* Receipt of nonstudy vaccines (with the exception of post-exposure vaccination in a medical emergency, eg, hepatitis, rabies, tetanus) within 3 weeks prior to Visit 1.
* Individuals who have ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.
* Individuals who have received antibiotics within 6 days before vaccination.
* Individuals with body temperature (axillary temperature) ≥38 degrees Celsius (≥ 100.4° F) within the last 3 days of intended study vaccination.
* BMI > 35 kg/m2.
* Female who are pregnant or nursing (breastfeeding) mothers or females of childbearing potential do not plan to use acceptable birth control measures, for the whole duration of the study. Adequate contraception is defined as hormonal (eg, oral, injection, transdermal patch, implant, cervical ring), barrier (eg, condom with spermicide or diaphragm with spermicide), intrauterine device (IUD), or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry; Abstinence.
* Individuals who are part of study personnel or close family members conducting this study.
* Individuals with history of substance or alcohol abuse within the past 2 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2902 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (25):
- Czechia (2):
  - Site 71 - Ordinace všeobecného lékaře, Kbel, Benátky Nad Jizerou
  - Site 70 - Vaccination and Travel Medicine Centre, Poliklinika II., Bratri Stefanu 895, Hradec Kralove
- Philippines (4):
  - Site 61 - Research Institute for Tropical Medicine DOH Compound, Filinvest Corporate City, Alabang Muntinlupa City
  - Site 60 - De La Salle Health Sciences Institute, Room 6210 and 6206 De La Salle Angelo King Medical Research Center, Congressional Road, Dasmarinas City, Cavite
  - Site 63 - Our Lady of Lourdes Hospital, 46 P. Sanchez Street, Sta., Mesa, Manila
  - Site 62 - Research Institute for Tropical Medicine DOH Compound, Filinvest Corporate City, Alabang, Muntinlupa City
- South Africa (15):
  - Site 33 - TREAD Research , Room 41, 8th Floor, Department of Cardiology, Tygerberg Hospital, Francie van Zijl Drive, Province of the Western Cape, Cape Town
  - Site 43 - Allergy Diagnostic & Clinical Research Unit, UCT Lung Institute, George Street, Province of the Western Cape, Cape Town
  - Site 34 - Synopsis Research, Room 8, First floor, Fountain Centre, Belmont Road, Rondebosch, Cape Town
  - Site 41 - Tiervlei Trial Centre, Karl Bremer Hospital, c/o Mike Pienaar Boulevard & Frans Conradie Avenue, Bellville, Western Cape, Cape Town
  - Site 45 - 343 Randles Road, Sydenham, Durban
  - Site 44 - Dr B van der Berg and Associates, 162 Pretoria Road, Rynfield, Benoni, Gauteng
  - Site 31 - MD Search, 1 Paul Smit Street, Boksburg North, Gauteng
  - Site 32 - EMMED Research, Emmed Research, 641 5th Avenue, Eloffsdal, Gauteng
  - Site 35 - I Engelbrecht Research (Pty) Ltd, 174 Cradock Avenue, Lyttleton, Gauteng
  - Site 36 - Midrand Medical Centre, Shop #1, Health Emporium, Cnr Church and Market Street, Midrand, Gauteng
  - Site 38 - Perinatal HIV Research Unit, New Nurses Home, Chris Hani Baragwanath Academic Hospital, Chris Hani Road, Soweto, Gauteng
  - Site 39 - Medicross Sophiatown, Cnr Edward and Millar Streets, Vrededorp, Gauteng
  - Site 37 - Excellentis Clinical Trial Consultants, Suite 201, York Building, 72, York Street, George
  - Site 40 - Newtown Clinical Research Centre, Suite 3, Newgate Centre, 104 Jeppe Street, Newtown, Johannesburg
  - Site 46 - Helderberg Clinical Trials Centre, Suite 7G&H Arun Place, Sir Lowry's Pass Road, Somerset West
- Thailand (4):
  - Site 53 - Clinical Trials Unit, Office for Research and Development, His Majesty the King's 80th Birthday December 2007 Building, 3rd floor, room 307, Faculty of Medicine Siriraj Hospital, Mahidol University, 2 Prannok Rd., Bangkoknoi, Bangkok
  - Site 52 - 1. Faculty of Medicine, Chulalongkorn University, Rama 4 Rd., Pathumwan, Bangkok
  - Site 52 - 2. Queen Saovabha Memorial Institute, Thai Red Cross Society, Rama 4 Rd., Pathumwan, Bangkok
  - Site 51 - Faculty of Medicine, Srinakharinwirot University, HRH Princess, Sirindhorn Medical Center, Ongkarak, Nakhorn, Nayok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 sites with 3 sites in Thailand, 4 sites in Philippines, 15 sites in South Africa and 2 sites in Czech Republic.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Agriflu: Subjects ≥50 years of age who received one vaccination of an investigational vaccine TIV
- Fluvirin: Subjects ≥50 years of age who received one vaccination of a control vaccine TIVf
Period: Overall Study
Arm/Group | Agriflu | Fluvirin
Started | 1452 | 1450
Completed | 1450 | 1440
Not Completed | 2 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Not Eligible | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Agriflu | Fluvirin | Total
Number analyzed (Participants) | 1452 | 1450 | 2902
Age, Continuous [Mean (Standard Deviation); unit: year] | 64.2 (8.9) | 64.2 (8.9) | 64.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 943 | 893 | 1836
  Male | 509 | 557 | 1066

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Geometric Mean Titers (GMTs) of TIV Group and TIVf Group for All Three Strains, in Healthy Adults Aged ≥50 Years
Description: Non-inferiority of Postvaccination Hemagglutination Inhibition (HI) Geometric Mean Titers (GMTs) of TIV (Trivalent Subunit Inactivated Influenza Vaccine) Group Over the Corresponding TIVf Group for All Three Strains, three weeks after vaccination (day 22).
  The upper limit of the two-sided 95% confidence interval (CI) on the ratio of GMTs (GMT TIVf/GMT TIV) should not exceed the non-inferiority margin of 1.5.
Time Frame: Day 22
Population: Analysis was done on the per-protocol set 1 (PPS1) , ie, the subjects who received the vaccine correctly; provided evaluable serum samples at visit 2; and had no major protocol violations as defined prior to analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Agriflu | Fluvirin
Number analyzed (Participants) | 1402 | 1397
Titers
  A/H1N1(1401, 1397) | 315 [281 to 352] | 581 [519 to 651]
  A/H3N2(1401, 1397) | 697 [635 to 764] | 1048 [955 to 1149]
  B | 36 [33 to 39] | 36 [33 to 39]
Statistical Analysis 1: Comparison: Agriflu vs Fluvirin; Non-inferiority of HI GMTs of TIV vaccine over HI GMTs of TIVf vaccine for the strain A/H1N1 at day 22; Test type: Non-Inferiority or Equivalence — The HI GMTs of TIV vaccine for strain A/H1N1 considered non-inferior to HI GMTs of TIVf vaccine if the upper limit of the two-sided 95% CI on the ratio of GMTs (GMT TIVf / GMT TIV) was ≤1.5; ANCOVA; Not applicable(NA); Ratio of GMTs = 1.85, 95% CI 2-sided [1.66 to 2.06]
Statistical Analysis 2: Comparison: Agriflu vs Fluvirin; Non-inferiority of HI GMTs of TIV vaccine over HI GMTs of TIVf vaccine for the strain A/H3N2 at day 22; Test type: Non-Inferiority or Equivalence — The HI GMTs of TIV vaccine for strain A/H3N2 considered non-inferior to HI GMTs of TIVf vaccine if the upper limit of the two-sided 95% CI on the ratio of GMTs (GMT TIVf / GMT TIV) was ≤1.5; ANCOVA; Ratio of GMTs = 1.5, 95% CI 2-sided [1.38 to 1.64]
Statistical Analysis 3: Comparison: Agriflu vs Fluvirin; Non-inferiority of HI GMTs of TIV vaccine over HI GMTs of TIVf vaccine for the strain B at day 22; Test type: Non-Inferiority or Equivalence — The HI GMTs of TIV vaccine for strain B considered non-inferior to HI GMTs of TIVf vaccine if the upper limit of the two-sided 95% CI on the ratio of GMTs (GMT TIVf / GMT TIV) was ≤1.5; ANCOVA; Ratio of GMTs = 1, 95% CI 2-sided [0.93 to 1.08]

2. Primary Outcome: Percentages of Subjects Achieving Seroconversion (SC) in Antibody Titers in the TIV Group Compared With the Corresponding Percentages of Subjects in the TIVf Group for All Three Strains At Day 22, in Healthy Adults Aged ≥50 Years
Description: Non-Inferiority was measured as the percentages of subjects who achieved seroconversion in HI titers three weeks (day 22) after vaccination of TIV compared with TIVf, against each of three vaccine strains.
  Seroconversion is defined as a prevaccination titer <10 and postvaccination HI ≥40 or as a prevaccination titer ≥10 and at minimum four-fold rise in postvaccination antibody titer.
  The upper limit of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion TIVf - SeroconversionTIV) should not exceed 10%.
Time Frame: Day 22
Population: Analysis was done on the PPS2, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at visit 1 and visit 2; and had no major protocol violations as defined prior to analysis
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Agriflu | Fluvirin
Number analyzed (Participants) | 1399 | 1391
percentages of subjects
  A/H1N1(1397,1391) | 75 [73 to 78] | 84 [82 to 86]
  A/H3N2(1398,1390) | 72 [70 to 74] | 85 [83 to 87]
  B(1399,1390) | 41 [39 to 44] | 40 [37 to 43]
Statistical Analysis 1: Comparison: Agriflu vs Fluvirin; Non-inferiority of percentage of subjects with HI seroconversion of TIV vaccine over TIVf vaccine for the strain A/H1N1 at day 22; Test type: Non-Inferiority or Equivalence — Percentage of subjects with HI seroconversion of TIV vaccine for strain A/H1N1 considered non-inferior to percentage of subjects with HI seroconversion of TIVf vaccine if the upper limit of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion TIVf - Seroconversion TIV) was ≤10%; Miettinen and Nurminen; Difference in seroconversion rates = 9, 95% CI 2-sided [5.6 to 11.5]
Statistical Analysis 2: Comparison: Agriflu vs Fluvirin; Non-inferiority of percentage of subjects with HI seroconversion of TIV vaccine over TIVf vaccine for the strain A/H3N2 at day 22; Test type: Non-Inferiority or Equivalence — Percentage of subjects with HI seroconversion of TIV vaccine for strain A/H3N2 considered non-inferior to percentage of subjects with HI seroconversion of TIVf vaccine if the upper limit of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion TIVf - Seroconversion TIV) was ≤10%; Miettinen and Nurminen; Difference in seroconversion rates = 13, 95% CI 2-sided [10.1 to 16.1]
Statistical Analysis 3: Comparison: Agriflu vs Fluvirin; Non-inferiority of percentage of subjects with HI seroconversion of TIV vaccine over TIVf vaccine for the strain B at day 22; Test type: Non-Inferiority or Equivalence — Percentage of subjects with HI seroconversion of TIV vaccine for strain B considered non-inferior to percentage of subjects with HI seroconversion of TIVf vaccine if the upper limit of the two-sided 95% CI on the difference between the seroconversion rates (Seroconversion TIVf - Seroconversion TIV) was ≤10%; Miettinen and Nurminen; Difference in seroconversion rates = -1, 95% CI 2-sided [-5 to 2.3]

3. Secondary Outcome: Evaluation of Percentages of Subjects Who Achieved HI Seroconversion and HI Titer ≥1:40 Against Each of Three Strains After One Vaccination of TIV and TIVf Vaccine
Description: Percentage of subjects achieving HI seroconversion against each of three vaccine strains was measured three weeks after vaccination of TIV and TIVf vaccine (day 22).
  Percentage of subjects who achieved HI titer ≥1:40 against each of three vaccine strains was measured three weeks after one vaccination of TIV and TIVf vaccine.
  According to Center for Biologics Evaluation and Research recommendations (CBER 2007), the criterion for seroconversion is considered met if the lower limit of the two-sided 95% CI for the percentage of subjects with HI seroconversion is ≥40% (<65 years) or ≥30% (≥65 years).
  As per the CBER criteria, the lower limit of the two-sided 95% CI for the percentage of subjects who achieved HI titer ≥ 1:40 should be ≥70% (<65 years) or ≥60% (≥65 years).
Time Frame: Day 22
Population: Analysis was done on the PPS1 for HI Titer ≥1:40 at day 22 and PPS2 for Seroconversion
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- ≥50 to ≤64 years_Agriflu: Subjects ≥50 to ≤64 years of age who received an investigational vaccine TIV
- ≥50 to ≤64 years_Fluvirin: Subjects ≥50 to ≤64 years of age who received a control vaccine TIVf
- ≥65 years_Agriflu: Subjects ≥65 years of age who received an investigational vaccine TIV
- ≥65 years_Fluvirin: Subjects ≥65 years of age who received a control vaccine TIVf
Arm/Group | ≥50 to ≤64 years_Agriflu | ≥50 to ≤64 years_Fluvirin | ≥65 years_Agriflu | ≥65 years_Fluvirin
Number analyzed (Participants) | 691 | 691 | 711 | 706
Percentages of subjects
  A/H1N1 - Seroconversion(687, 686, 710, 705) | 78 [74 to 81] | 87 [84 to 89] | 73 [70 to 77] | 81 [78 to 84]
  A/H3N2 - Seroconversion(688, 686, 710, 704) | 78 [75 to 81] | 88 [85 to 90] | 66 [63 to 70] | 82 [79 to 85]
  B - Seroconversion(688, 686, 711, 704) | 44 [40 to 48] | 45 [41 to 49] | 39 [35 to 42] | 35 [32 to 39]
  A/H1N1 - HI ≥1:40 (Day 22)[691, 691, 710, 706] | 94 [92 to 96] | 96 [94 to 97] | 91 [89 to 93] | 92 [90 to 94]
  A/H3N2 - HI ≥1:40 (Day 22)[691, 691, 710, 706] | 99 [99 to 100] | 99 [98 to 100] | 99 [98 to 99] | 98 [97 to 99]
  B - HI ≥1:40 (Day 22)[691, 691, 711, 706] | 58 [55 to 62] | 59 [55 to 63] | 59 [55 to 62] | 56 [52 to 60]

4. Secondary Outcome: Geometric Mean Ratio of Subjects Against Each of Three Strains After One Vaccination of TIV and TIVf Vaccine
Description: Geometric mean ratio (GMR) of subjects was calculated as the ratio of postvaccination to prevaccination HI GMTs against each of three vaccine strains, three weeks after vaccination of TIV and TIVf vaccine (day 22).
Time Frame: Day 22
Population: Analysis was done on the PPS1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | ≥50 to ≤64 years_Agriflu | ≥50 to ≤64 years_Fluvirin | ≥65 years_Agriflu | ≥65 years_Fluvirin
Number analyzed (Participants) | 688 | 686 | 711 | 705
Ratios
  A/H1N1(687, 686, 710, 705) | 18 [15 to 22] | 35 [29 to 42] | 15 [12 to 19] | 27 [21 to 33]
  A/H3N2(688, 686, 710, 704) | 13 [11 to 15] | 18 [15 to 20] | 9.65 [7.94 to 12] | 16 [13 to 20]
  B(688, 686, 711, 704) | 3.85 [3.43 to 4.31] | 3.91 [3.49 to 4.39] | 3.1 [2.71 to 3.54] | 3 [2.62 to 3.44]

5. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Adverse Events After One Vaccination of TIV and TIVf
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events from day 1 up to and including day 7 after vaccination of TIV and control.
Time Frame: Day 1 to 7 postvaccination
Population: Analysis was done on the safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Subjects
Arm/Group | Agriflu | Fluvirin
Number analyzed (Participants) | 1428 | 1433
Subjects
  Pain(1412, 1424) | 264 | 254
  Ecchymosis Type I(1419, 1425) | 26 | 33
  Ecchymosis Type II(1419, 1425) | 7 | 11
  Erythema Type I(1410, 1427) | 91 | 93
  Erythema Type II(1410, 1427) | 16 | 10
  Induration Type I(1423, 1429) | 78 | 65
  Induration Type II(1423, 1429) | 25 | 19
  Swelling Type I(1419, 1427) | 50 | 44
  Swelling Type II(1419, 1427) | 21 | 15
  Chills(1403,1407) | 64 | 68
  Malaise(1402,1405) | 88 | 95
  Nausea(1401,1405) | 48 | 44
  Myalgia(1400,1403) | 128 | 140
  Arthralgia(1396,1403) | 83 | 87
  Headache(1397,1403) | 153 | 161
  Sweating(1403,1405) | 99 | 102
  Fatigue(1404,1407) | 143 | 145
  Loss of Appetite(1404,1403) | 43 | 59
  Fever(>=38°C)[1422,1428] | 20 | 21

ADVERSE EVENTS:
Time Frame: Up to 22 days
Description: Adverse events and Serious Adverse Events were collected from day 1 through day 22.
  The number of subjects analyzed in this section is from the safety set. Safety Set (Overall) includes all subjects in the exposed set who had either postvaccination AE or solicited AE data.
Groups:
- Total: Total number of Subjects
Arm/Group | Agriflu | Fluvirin | Total
Serious Adverse Events (participants affected / at risk) | 3/1452 | 5/1445 | 8/2897
Other Adverse Events (participants affected / at risk) | 471/1452 | 467/1445 | 938/2897
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agriflu (N=1452) | Fluvirin (N=1445) | Total (N=2897)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1 | 2
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 1
HYPERTENSION (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Agriflu (N=1452) | Fluvirin (N=1445) | Total (N=2897)
Fatigue (General disorders) | 144 | 146 | 290
Injection Site Pain (General disorders) | 281 | 276 | 557
Malaise (General disorders) | 89 | 95 | 184
Arthralgia (Musculoskeletal and connective tissue disorders) | 85 | 88 | 173
Myalgia (Musculoskeletal and connective tissue disorders) | 133 | 141 | 274
Headach (Musculoskeletal and connective tissue disorders) | 159 | 164 | 323
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 99 | 103 | 202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial